#### IRB -TPEVGH SOP 05-01 附表 4-1

Version: 2.0, Date: 2015/06/16

# 臺北榮民總醫院人體試驗委員會臨床試驗計畫中文計畫書摘要

- 一、計畫名稱:運用動物輔療於護理之家改善住民之認知及情緒
- 二、計畫主持人、醫師、研究人員及試驗進行地點:

計畫主持人:王素貞護理師

共同主持人: 鄒芳榆護理長、林沂螢副護理長

試驗進行地點:臺北榮民總醫院桃園分院附設松柏園護理之家

## 三、研究背景:

於臺灣之護理安養機構有收治失智症之住民,在照顧上常有精神及情緒問題,使用藥物來改善住民的精神及情緒狀況是常見之措施;現多有研究將非藥物治療如:園藝、懷舊、寵物…等等不同介入措施於失智長者,皆有成效;針對治療犬方面,治療犬與治療犬帶領員經過一系列訓練,社會化後與人親近,透過指令與人進一步互動;國內研究觀察多位失智者於有活動有寵物治療非藥物介入措施的研究中,寵物治療能改善失智症的照護品質,減少精神方面不適切的藥物使用,並延緩退化。國外研究針對失智症的安養機構住民安排每週一次與治療犬一起活動的介入措施,為期 6 個月,結果是安養機構住民於社交互動、情緒表達以及行為和心理症狀皆有益的明顯改善。

本家護理機構有八成多為失智症之住民,於精神及情緒上常有不穩定之狀況,相對影響工作人員及照服員需花時間協助排除問題;希望可以加入非藥物介入措施,如寵物治療,期望能改善失智症的精神及情緒不適切表現,減少干擾行為,使住民之生活照護品質改善,進一步能減少精神方面不適切的藥物使用,期許住民於生理機能上延緩退化。

## 四、研究目的:

主要目的:安排治療犬與護理之家住民互動,雖非侵入性介入措施,但有因聽覺、視覺及觸覺上之感受,期望藉由量化之評估,可以改善生活功能、認知狀態及情緒。

次要目的:期望質性上可以觀察住民情緒穩定,夜眠佳,增加社 交互動之行為。

## 五、研究步驟:

- (一)介入措施:12 週 30~40 分鐘安排課程使住民與治療犬互動。
- (二)研究工具:運用自構式調查表、巴氏量表(Barthel index)、

#### PRB-TPEVGH SOP 05-01 附表 4-1

Version: 2.0, Date: 2015/06/16

簡短智能問卷 (Short Portable mental state questionnaire 簡稱 SPMSQ), 老年憂鬱症量表(GDS)及簡式健康量表(心情溫度計)。

- 1. 自構式調查表包括病患基本屬性。
- 2. 巴氏量表(Barthel index) 了解住民之日常生活功能。
- 3. 認知方面使用簡短智能問卷 (Short Portable mental state questionnaire 簡稱 SPMSQ)評估
- 4. 使用老年憂鬱症量表(GDS)及簡式健康量表(心情溫度計)來檢 視住民之情緒狀況。
- (三)收案流程:介入措施前先收集自構式調查表、巴氏量表 (Barthel index)、簡短智能問卷 (Short Portable mental state questionnaire 簡稱 SPMSQ)、老年憂鬱症量表(GDS)及簡式健康量表(心情溫度計)。
- 1. 實驗組:安排每週一次介入措施, 共接受 12 次介入措施。
- 2. 對照組: 與實驗組同日同時段安排每週一次一般照護活動,共 12次。
- 3. 於執行開始後第8週、12週、16週時再進行第2~4次評估巴氏量表(Barthel index)、簡短智能問卷 (Short Portable mental state questionnaire 簡稱 SPMSQ)、老年憂鬱症量表 (GDS)及簡式健康量表(心情溫度計)

## 六、研究設計:

- 1. 進行方式:實驗性平行之研究設計。
- 2. 是否有對照組:有。
- 3. 盲化方式:單盲。
- 4. 隨機分派:是隨機分派;接受介入措施之實驗組與一般常規照 護之對照組的評估,採前後測進行資料收集。採簡單隨機分 派方式,收案單號為實驗組,收案雙號對照組。

# 七、受試者:

- 納入標準:為本護理之家之住民,住民或家屬意識清楚,可 國台語溝通,住民無對犬類過敏、攻擊、排斥、不舒服之 感受,說明研究流程及同意參與並簽署同意書者。
- 排除標準:住民無法配合者,對犬類有過敏、攻擊、排斥、 不舒服之感受,篩選後不適合、不同意簽署受試者同意書

#### **BRB-TPEVGH SOP 05-01 附表 4-1**

Version: 2.0, Date: 2015/06/16

竿。

## 3. 受試者數目:

受試者數目及計算以 G-POWER 3.1.9.7 版軟體進行計算,test family: F-tests,statistical test: ANOVA: Repeated measures, within-between interaction,Type of power analysis: A priori: Compute required sample size-given  $\alpha$ , power, and effect size. Effect size: 0.20,  $\alpha$  error: 0.05, power( $1-\beta$  error): 0.8, number of groups: 2, number of measurements: 4, 樣本數共 36 人,實際效力: 0.80。但實際上收集資料可能遭遇到的困難,或病情變化而不想參與研究等等,因而減少收案數,故預估流失率約 10~15%,預計收案約 40~42 人,實驗組及對照組各 20~21 人。

## 八、研究方法

- 1. 介入措施治療程序:介入措施為安排課程使住民與治療犬互動,每週一次30~40分鐘、治療期共12週。
- 2. 試驗期間的併用療法:無。
- 3. 試驗所要做之臨床觀察:量性方面數據巴氏量表(Barthel index)、簡短智能問卷 (Short Portable mental state questionnaire 簡稱 SPMSQ),老年憂鬱症量表(GDS)及簡式健康量表(心情溫度計)。
- 4. 追蹤時間表:於執行開始後第8週、12週、16週時再進行第 2~4次評值,第16週追蹤後即停止追蹤。
- 5. 主要療效或評估指標:
  - (1) 臨床觀察是否改善住民生理及心理之生活品質,包括改善生活功能、延緩認知退化及穩定情緒狀態,來作為主要療效或評估指標。
  - (2) 療效判定標準量性數據 p<0.05 為有效。

### 九、副作用處理

1. 副作用標準及發生率:治療犬經過社會化訓練,情緒穩定及 聽從指令,並有健康及定期施打疫苗證明;對受試者或家 屬說明研究內容前,先了解住民有無對犬類過敏、攻擊、 排斥、不舒服之感受,如沒有者才納入受試者,但副作用 如因研究執行過程有不舒服、過敏或情緒欠穩等,其發生 機率應屬少數狀況,無法估計發生率。

#### 4RB-TPEVGH SOP 05-01 附表 4-1

Version: 2.0, Date: 2015/06/16

- 回報方式:因研究人員於現場,當研究對象有副作用發生時, 應立即回報研究主持人。
- 3. 處理方式:副作用發生時,如是情緒狀態,可暫帶離現場給 予安撫如有加劇,可掛精神科身心門診,如有皮膚過敏可 皮膚科門診求治,如有生命徵象欠穩則送急診臺北榮民總 醫院桃園分院求治;以上副作用皆需聯繫個案之家屬及說 明。

## 十、 受試者權益

- 1. 隱私保護:收案前經由研究人員向所有受試者或家屬說明研究流程,進行知情同意的場所,於護理之家之會客室,以避免被他人旁觀或旁聽,不影響治療及醫囑,簽署同意書後才開始進行研究,過程中隨時可退出研究。填寫完畢的資料只做學術研究使用,不做另外其他用途,並不會公布參與者生名。研究資料保密方面:保存文件或檔案之櫃子須上鎖,盡量以編碼代替可辨識身分之資料,並妥為保存編碼表,儲存檔案之電腦、隨身碟、外接硬碟等設備,設定開機密碼;設定受試者資料的使用人權限,儘量減少使用可攜式儲存設備,例如筆電、隨身碟、外接硬碟等,也盡量避免使用 E-mail 傳送含有個資之檔案。
- 2. 倫理問題:基於保護參與研究的人類受試者之倫理原則 (principles)與指引(guidelines),貝爾蒙原則(Belmont principles)本的倫理考量。對於研究對象需尊重人格 (respect for persons)之原則,保障參與者的自主性、知情 同意、隱私與資料保密、必須對自主性較低者提供特別保護。 依行善(beneficence)原則上,考量研究設計之適當性、對可 能風險是否提供安全上或防護的措施、預期之利益與風險是 否有適當的比例、是否將使風險減少至最小化等。依正義 (iustice)原則上,考量研究收案對象的標準是否有符合正 義、研究結果與負擔之分配是否有公平、其個人或族群是否 可從研究結果中獲得益處等等考量。此研究與過程根據臺北 榮民總醫之人體研究案件範圍檢核,雖有設計非侵入性之介 入措施,但是研究內容為個人或群體特質或行為,但不含造 成個人或族群歧視之潛在可能者,根據本實驗之研究設計易 取樣,因對象為易受傷之族群(無法自主行使同意之成人、經 濟弱勢或教育弱勢者),故送一般審查。研究倫理方面,身為 嚴謹的研究者須要了解與學習,人權之重要性永遠在科學之

#### **FRB-TPEVGH SOP 05-01 附表 4-1**

Version: 2.0, Date: 2015/06/16

上,研究科學的態度是謙卑地,對於研究對象必須給予平等及尊重。

3. 遵守不傷害原則:執行介入性活動時,計畫主持人或共同主持人皆會在場協助,若受試者有感受不適或中途想退出,可隨時停止資料的收集,避免對受試者造成心理的創傷,給予陪伴與心理支持,必要時轉介給收案醫院(臺北榮民總醫院桃園分院)的社工師或身心科門診,給予心理輔導及精神諮詢。

## 十一、統計分析

- 1. 描述統計:分析基本屬性之類別資料以人數、次數與百分比 呈現,連續資料以最大值、最小值、百分比、平均 數與標準差呈現;卡方檢定兩組同質性。
- 2. 推論統計:以卡方檢定兩組類別變項、以 t-test 檢定兩組連續變項;重複測量以廣義估計方程式(Generalized estimating equations, GEE)分析來檢定主要介入措施的療效指標成效。
- 3. 期間分析:無進行期間分析,待收齊四次資料後再進行分析。 十二、附錄